CLINICAL TRIAL: NCT06520995
Title: The Effect of Education Program Supported by Cognitive Exercises in Elderly Individuals With Type 2 Diabetes
Brief Title: Elderly Patients With Type 2 Diabetes and Cognitive Exercises
Acronym: DIACOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hande Bulut Canbaz, RN, Msc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/183
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Impairment; Diabetes Mellitus, Type 2; Diabetes Complications
MeSH Terms: conditions — Cognitive Dysfunction; Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Patients in this group will only receive standard diabetes education.
- Video Group (Experimental): In addition to standard diabetes education, patients in this group will be educated with the mentioned video education program (a total of 12 diabetes education videos prepared by the researcher).
  Interventions: Other: Educational video program
- Video and Mobile application Group (Experimental): In addition to standard diabetes education and video education, patients in this group will participate in cognitive exercises for 15-20 minutes a day for 3 months via a mobile application.
  Interventions: Other: Educational video program; Other: A mobile application

INTERVENTIONS:
Other: Educational video program — Diabetes education video contents are as follows; Type 2 diabetes definition, symptoms and the effect of diabetes on cognitive functions, Medical nutrition therapy and healthy nutrition recommendations in Type 2 diabetes, The importance of diabetes and exercise, Oral antidiabetic treatments, Insulin treatment, Hypoglycemia symptoms, findings and treatment, Macrovascular complications in diabetes, Microvascular complications in diabetes, Foot Protection and care recommendations, Diabetes self-care skills and problem-solving strategies, Diabetes and stress management.
  Arms: Video Group; Video and Mobile application Group
Other: A mobile application — This mobile application is a science-based application that patients can access via their smartphone or tablet. It consists of verbal, numerical, visual, logical, memory and attention categories and contains 24 different gamified mind exercises
  Arms: Video and Mobile application Group

SUMMARY:
The study was planned as a single-center, prospective randomized controlled study. Individuals over 65 years of age with type 2 diabetes without severe cognitive impairment will be included in the study. The primary aim of the study is to improve the cognitive functions of the patients after the interventions. The secondary aim is to strengthen patients' diabetes self-management and increase their quality of life, especially by improving their glycemic control. For these purposes, in our study, patients will be randomized into three groups: "cognitive exercise and diabetes education", "diabetes education only" and "control" group. The control group will be provided with standard outpatient diabetes education. Individuals who will be in the "cognitive exercise and video training" group will watch a total of 12 diabetes education videos prepared by the researcher, in which a different topic will be discussed every week for 3 months, and they will also participate cognitive exercises for 15-20 minutes a day for 3 months via a mobile application. Individuals in the "diabetes education only" group will similarly watch a total of 12 diabetes education videos prepared by the researchers. Patients will be evaluated in terms of cognitive function, psychosocial problems (anxiety, depression, stress), glycemic control (HbA1c), diabetes management and quality of life before the interventions, at 3 months and 6 months.

DETAILED DESCRIPTION:
The aim of this study is to strengthen patient outcomes and diabetes management in individuals with diabetes through cognitive-based diabetes education. The study was planned as a single-center, prospective randomized controlled study. İndividuals over 65 years of age with type 2 diabetes with without severe cognitive impairment will be included in the study. In the study, patients will receive diabetes education and cognitive exercise for 12 weeks. In the study, patients will be randomized into three groups: "cognitive exercise and diabetes education", "diabetes education only" and "control" group. The control group will be provided with standard outpatient diabetes education. Patients will be evaluated in terms of cognitive function, psychosocial problems (anxiety, depression, stress), glycemic control (HbA1c), diabetes management and quality of life before the interventions, at 3 months and 6 months.

In the study, diabetes education will be provided through short, understandable diabetes education videos prepared by the researcher with up-to-date guide information. A total of 12 videos will be sent to patients' phones, covering a different topic each week for 3 months. Diabetes education video contents are as follows; Type 2 diabetes definition, symptoms and the effect of diabetes on cognitive functions, Medical nutrition therapy and healthy nutrition recommendations in Type 2 diabetes, The importance of diabetes and exercise, Oral antidiabetic treatments, Insulin treatment, Hypoglycemia symptoms, findings and treatment, Macrovascular complications in diabetes, Microvascular complications in diabetes, Foot Protection and care recommendations, Diabetes self-care skills and problem-solving strategies, Diabetes and stress management.

A mobile application will be used as a cognitive exercise tool in the study. This mobile application is a science-based application that patients can access via their smartphone or tablet. It consists of verbal, numerical, visual, logical, memory and attention categories and contains 24 different gamified mind exercises.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least one year
* Literate
* Able to use smartphone/tablet/computer and have internet access
* Individuals who agree to participate in the study will be included.

Exclusion Criteria:

* Type 1 diabetes
* With severe cognitive impairment
* Known neurological or psychiatric disorders
* Severely depressed
* Individuals with disabilities (vision, hearing problems, etc.) will not be included in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive profile | The moment it is included in the study, 3rd month, 6th month
  Neurocognitive Assessment Battery

SECONDARY OUTCOMES:
Hba1c | The moment it is included in the study, 3rd month, 6th month
  Laboratory values derived from patients' routine visits
Psychological state | The moment it is included in the study, 3rd month, 6th month
  A Scale to assess psychological state
Quality of Life (1) | The moment it is included in the study, 3rd month, 6th month
  Burden of Diabetes in the Elderly Scale
Quality of Life (2) | The moment it is included in the study, 3rd month, 6th month
  Type 2 Diabetes Self-Management Scale
Qality of Life (3) | The moment it is included in the study, 3rd month, 6th month
  SF-12 Quality of Life Scale
Cognitive Function (2) | The moment it is included in the study, 3rd month, 6th month
  Cognitive Function Instrument-Participant Form

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Tulek, RN,Prof. Dr., Study Director — Istanbul University-Cerrahpasa, Florence Nightingale Faculty of Nursing; Hande Bulut Canbaz, RN,Msc, Principal Investigator — Istanbul University-Cerrahpasa, Florence Nightingale Faculty of Nursing
Locations (1):
- Istanbul University-Cerrahpasa, Florence Nightingale Faculty of Nursing, Istanbul, Avcılar, Turkey (Türkiye)